CLINICAL TRIAL: NCT04975477
Title: CHESS-SAVE Score to Stratify Decompensation Risk in Compensated Advanced Chronic Liver Disease: an International Multicenter Study (CHESS2102)
Brief Title: CHESS-SAVE Score to Stratify Decompensation Risk in Compensated Advanced Chronic Liver Disease (CHESS2102)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Collaborators: LanZhou University (Other); Institute of Liver and Biliary Sciences (ILBS) (Unknown); Zagazig University (Other Government); Korea University (Other); Ehime University Graduate School of Medicine (Other); Hyogo Medical University (Other); Tianjin Second People's Hospital (Other); Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Xiaolong Qi, Chief, Hepatopancreatobiliary Surgery Institute of Gansu Province
Other Study IDs: CHESS2102
Record Dates: First submitted 2021-07-14; First posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Compensated Advanced Chronic Liver Disease
Keywords: liver stiffness; platelets; albumin; varices; compensated cirrhosis
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Training cohort: A cohort was used to develop the novel score for predicting liver decompensation
  Interventions: Procedure: Esophagogasrtoduodendoscopy and liver stiffness
- Validation cohort: A cohort was used to validate the performance of novel score for predicting liver decompensation
  Interventions: Procedure: Esophagogasrtoduodendoscopy and liver stiffness
- Exploratory cohort: A cohort was used to study the diagnostic value of novel score for clinically significant portal hypertension
  Interventions: Procedure: Esophagogasrtoduodendoscopy and liver stiffness; Procedure: hepatic venous pressure gradient

INTERVENTIONS:
Procedure: Esophagogasrtoduodendoscopy and liver stiffness — Time frame between elastography measurement and esophagogastroduodendoscopy is within 6 months.
Procedure: hepatic venous pressure gradient — A method was used to evaluate portal pressure.
  Groups: Exploratory cohort

SUMMARY:
Compensated advanced chronic liver disease (cACLD) was associated with a high rate of variceal bleeding, ascites, and hepatic encephalopathy due to portal hypertension. In these patients, esophagogastroduodenoscopy and hepatic venous pressure gradient were recommended methods to evaluate portal hypertension. However, non-invasive predictors of outcomes to stratify care remains needed. Although the updated EASL guideline has recommended that patients with liver stiffness >20kPa or platelets <150*10^9/L had the high risk of decompensation, the criteria remains to be validated. This international multicenter study aims to develop a novel CHESS-SAVE score to further predict the risk of liver decompensation in cACLD patients.

DETAILED DESCRIPTION:
Compensated advanced chronic liver disease (cACLD) was associated with a high rate of variceal bleeding, ascites, and hepatic encephalopathy due to portal hypertension. In these patients, esophagogastroduodenoscopy and hepatic venous pressure gradient were recommended methods to evaluate portal hypertension. However, non-invasive predictors of outcomes to stratify care remains needed. Although the updated EASL guideline has recommended that patients with liver stiffness >20kPa or platelets <150*10^9/L had the high risk of decompensation, the criteria remains to be validated. This international multicenter study initialed and enrolled by Chinese Portal Hypertension Alliance (CHESS) aims to develop a novel CHESS-SAVE score to further predict the risk of liver decompensation in cACLD patients.

ELIGIBILITY:
Training and validation cohort

Inclusion Criteria:

* age more than 18 years;
* fulfilled diagnosis of cACLD based on radiological, histological features of liver cirrhosis

Exclusion Criteria:

* prior liver decompensation;
* hepatocellular carcinoma;
* prior liver transplantation;
* portal vein thrombosis;
* antiplatelet or anticoagulation;
* without screening EGD within six months of TE;
* incomplete follow-up data.

HVPG cohort

Inclusion Criteria:

* age more than 18 years;
* fulfilled diagnosis of cACLD based on radiological, histological features of liver cirrhosis

Exclusion Criteria:

* prior liver decompensation;
* hepatocellular carcinoma;
* prior liver transplantation;
* portal vein thrombosis;
* antiplatelet or anticoagulation;
* without screening EGD within six months of TE;
* without HVPG measurement;
* non-sinusoidal portal hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients were fulfilled diagnosis of cACLD based on radiological, histological features of liver cirrhosis.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-07-16 (Estimated); Primary Completion 2021-08-16 (Estimated); Study Completion 2021-08-16 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the CHESS-SAVE score for predicting liver decompensation | 3 years
  To assess the accuracy of the CHESS-SAVE score to predict liver decompensation in patients with compensated advanced chronic liver disease

CONTACTS AND LOCATIONS:
Locations (7):
- China (2):
  - Ruijin Hospital, Shanghai
  - Tianjin Second People's Hospital, Tianjin
- Zagazig University Faculty of Medicine, Zagazig, Egypt
- Institute of Liver and Biliary Sciences, New Delhi, India
- Japan (2):
  - Ehime University Graduate School of Medicine, Matsuyama
  - Hyogo College of Medicine, Nishinomiya
- Korea University Ansan Hospital, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Qi X, Berzigotti A, Cardenas A, Sarin SK. Emerging non-invasive approaches for diagnosis and monitoring of portal hypertension. Lancet Gastroenterol Hepatol. 2018 Oct;3(10):708-719. doi: 10.1016/S2468-1253(18)30232-2. PMID 30215362
- [Background] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Background] Villanueva C, Albillos A, Genesca J, Garcia-Pagan JC, Calleja JL, Aracil C, Banares R, Morillas RM, Poca M, Penas B, Augustin S, Abraldes JG, Alvarado E, Torres F, Bosch J. beta blockers to prevent decompensation of cirrhosis in patients with clinically significant portal hypertension (PREDESCI): a randomised, double-blind, placebo-controlled, multicentre trial. Lancet. 2019 Apr 20;393(10181):1597-1608. doi: 10.1016/S0140-6736(18)31875-0. Epub 2019 Mar 22. PMID 30910320
- [Background] Sarin SK, Lamba GS, Kumar M, Misra A, Murthy NS. Comparison of endoscopic ligation and propranolol for the primary prevention of variceal bleeding. N Engl J Med. 1999 Apr 1;340(13):988-93. doi: 10.1056/NEJM199904013401302. PMID 10099140
- [Background] Cholongitas E, Papatheodoridis GV, Vangeli M, Terreni N, Patch D, Burroughs AK. Systematic review: The model for end-stage liver disease--should it replace Child-Pugh's classification for assessing prognosis in cirrhosis? Aliment Pharmacol Ther. 2005 Dec;22(11-12):1079-89. doi: 10.1111/j.1365-2036.2005.02691.x. PMID 16305721
- [Background] Chen RC, Cai YJ, Wu JM, Wang XD, Song M, Wang YQ, Zheng MH, Chen YP, Lin Z, Shi KQ. Usefulness of albumin-bilirubin grade for evaluation of long-term prognosis for hepatitis B-related cirrhosis. J Viral Hepat. 2017 Mar;24(3):238-245. doi: 10.1111/jvh.12638. Epub 2016 Nov 14. PMID 27862671
- [Background] Abraldes JG, Bureau C, Stefanescu H, Augustin S, Ney M, Blasco H, Procopet B, Bosch J, Genesca J, Berzigotti A; Anticipate Investigators. Noninvasive tools and risk of clinically significant portal hypertension and varices in compensated cirrhosis: The "Anticipate" study. Hepatology. 2016 Dec;64(6):2173-2184. doi: 10.1002/hep.28824. Epub 2016 Oct 27. PMID 27639071
- [Background] Thabut D, Bureau C, Layese R, Bourcier V, Hammouche M, Cagnot C, Marcellin P, Guyader D, Pol S, Larrey D, De Ledinghen V, Ouzan D, Zoulim F, Roulot D, Tran A, Bronowicki JP, Zarski JP, Goria O, Cales P, Peron JM, Alric L, Bourliere M, Mathurin P, Blanc JF, Abergel A, Serfaty L, Mallat A, Grange JD, Attali P, Bacq Y, Wartelle-Bladou C, Dao T, Pilette C, Silvain C, Christidis C, Capron D, Bernard-Chabert B, Hillaire S, Di Martino V, Sutton A, Audureau E, Roudot-Thoraval F, Nahon P; ANRS CO12 CirVir group. Validation of Baveno VI Criteria for Screening and Surveillance of Esophageal Varices in Patients With Compensated Cirrhosis and a Sustained Response to Antiviral Therapy. Gastroenterology. 2019 Mar;156(4):997-1009.e5. doi: 10.1053/j.gastro.2018.11.053. Epub 2019 Feb 13. PMID 30768988
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines on non-invasive tests for evaluation of liver disease severity and prognosis - 2021 update. J Hepatol. 2021 Sep;75(3):659-689. doi: 10.1016/j.jhep.2021.05.025. Epub 2021 Jun 21. PMID 34166721
- [Derived] Liu C, Cao Z, Yan H, Wong YJ, Xie Q, Hirooka M, Enomoto H, Kim TH, Hanafy AS, Liu Y, Huang Y, Li X, Kang N, Koizumi Y, Hiasa Y, Nishimura T, Iijima H, Jung YK, Yim HJ, Guo Y, Zhang L, Ma J, Kumar M, Jindal A, Teh KB, Sarin SK, Qi X. A Novel SAVE Score to Stratify Decompensation Risk in Compensated Advanced Chronic Liver Disease (CHESS2102): An International Multicenter Cohort Study. Am J Gastroenterol. 2022 Oct 1;117(10):1605-1613. doi: 10.14309/ajg.0000000000001873. Epub 2022 Jun 15. PMID 35973168